CLINICAL TRIAL: NCT04358133
Title: Relieving Dyspnea With Low Dose of Morphine in Patients Admitted to the Intensive Care Unit for an Acute Respiratory Failure: a Double-blind Randomized Controlled Pilot Study
Brief Title: Low Dose Morphine to Relieve Dyspnea in Acute Respiratory Failure (OPIDYS)
Acronym: OPIDYS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRC18023; 2019-003091-39 (EudraCT Number)
Record Dates: First submitted 2020-03-31; First posted 2020-04-24 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Failure
Keywords: Acute respiratory failure; Dyspnea; Opioids; Comfort; Intensive care unit
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group,single center, phase 2 pilot study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The experimental group will receive an intravenous titration of morphine followed by a subcutaneous administration of morphine hydrochloride for 24 hours according to a predefined protocol. The control group will receive placebo NaCl 0.9% administered according to the same protocol as the experimental arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhydrate de morphine (Experimental): initial dose of 2 mg, followed by 1 mg every 3 minutes until a VAS-dyspnea <40 then relay subcut
  Interventions: Drug: Chlorhydrate de morphine
- NaCl 0,9% (Placebo Comparator): initial dose of 2 mg, followed by 1 mg every 3 minutes until a VAS-dyspnea <40 then relay subcut
  Interventions: Drug: NaCl 0,9%,

INTERVENTIONS:
Drug: Chlorhydrate de morphine — The experimental group will receive an intravenous titration of morphine followed by a subcutaneous administration of morphine hydrochloride for 24 hours according to a predefined protocol
  Arms: Chlorhydrate de morphine
Drug: NaCl 0,9%, — The control group will receive placebo NaCl 0.9% administered according to the same protocol as the experimental arm
  Arms: NaCl 0,9%

SUMMARY:
This study evaluates a pharmacological intervention to relieve dyspnea in intensive care unit patients. Indeed, opioids can be particularly beneficial since 1) dyspnea and pain share many similarities, 2) the benefit of opioids on dyspnea has been clearly demonstrated in other populations. However, to date, data regarding the impact of morphine on dyspnea in intensive care unit patients admitted for acute respiratory failure are scarce. There may be a reluctance of physicians to prescribe opioids that is not scientifically justified.

The study will focus on patient reported outcome (PRO) criteria. The ultimate goal of this pilot study is to design the protocol of a future pragmatic trial.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel-group, single-center phase 2 pilot study.The experimental group will receive an intravenous titration of morphine followed by a subcutaneous administration of morphine hydrochloride for 24 hours according to a predefined protocol. The control group will receive placebo NaCl 0.9% administered according to the same protocol as the experimental arm Patients will be randomized 1:1 between low-dose titrated morphine (experimental group) and placebo (control group). The other treatments will be similar in both groups, according to the protocol and the recommendations.

Severe dyspnea will be assessed for regularly Patients will be followed for 48 hours: 24-hour treatment duration, evaluation of primary endpoint for first 24 hours, collection of adverse events for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≤ 75 years
* Admitted in intensive care for an acute respiratory failure defined as a respiratory rate> 24 / min or signs of respiratory distress such as labored breathing or paradoxical inspiration, or SpO2 <90% in ambient air
* Spontaneous ventilation, either under standard oxygen, high flow oxygen or non invasive ventilation
* Dyspnea ≥ 40 on an dyspnea-VAS from zero (no dyspnea) to 100 (worst possible dyspnea)
* Richmond agitation and sedation scale (RASS) between 0 and 2.
* No confusion, as defined by the CAM-ICU
* Signed informed consent

Exclusion Criteria:

* Intubated patient
* Intubation planned upon admission
* Hearing or visual impairment
* Insufficient command of French
* Previous psychiatric or cognitive disorders known
* Moribund patient
* Known hypersensitivity to opioids
* Severe renal insufficiency (creatinine clearance <30 ml / min)
* Severe hepatocellular insufficiency (factor V <50%)
* Any formal contra-indication of opiates
* Opioid use within the 24 hours before inclusion
* Pregnancy or breastfeeding
* Minor and protected adult
* Exclusion period due to inclusion in another clinical trial
* Previous inclusion in this study
* No affiliation to social security

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Average dyspnea over 24 hours | systematically evaluated every 4 hours over 24 hours and whenever necessary
  Dyspnea will be assessed by VAS-dyspnea (ranging from zero, no dyspnea to 100, worst possible dyspnea) patient reported outcome criteria (PRO).

SECONDARY OUTCOMES:
Intensity of dyspnea | every 4 hours over 24 hours
  patient reported outcome measure (PRO) ; min=0;max=100(worse)
Incidence of severe dyspnea (dyspnea ≥40) | within 24 hours
  patient reported outcome measure (PRO) ; min=0;max=100(worse)
Anxiety | every 4 hours as well as over the first 24 hours
  Patient reported outcome measure (PRO) ; min=0;max=100(worse)
Incidence of moderate to severe anxiety | every 4 hours over 24 hours
  Incidence of moderate to severe anxiety (PRO) ; min=0;max=100(worse)
Intubation rate | within the first 48 hours
  Intubation rate
Vigilance level (Glasgow Coma Scale : impaired alertness defined by Glasgow Coma Scale ≤ 12) | every 4 hours as well as the first 48 hours
  Vigilance level ; GCS : min=3(worse) ;max=15
Incidence of coma | within the first 48 hours
  Incidence of coma
Incidence of delirium | within the first every 4 hours as well as over the first 48 hours
  Incidence of delirium
Respiratory rate | every 4 hours as well as over the first 24 hours
  Respiratory rate
Proportion of patients requiring the transition from one oxygenation technique to another | At the end of the study (12 months)
  Proportion of patients requiring the transition from one oxygenation technique to another
Intensity of pain | every 4 hours
  Patient reported outcome measure (PRO) ; min=0;max=100(worse)
Duration of night sleep the first night | at the end of the first night
  Duration of night sleep the first night (number of hours)
Quality of sleep the first night | at the end of the first night
  Patient reported outcome measure (PRO); min=0;max=100(worse)
Severity of dry eye | in the first 24 hours
  Patient reported outcome criteria (PRO); min=0;max=100(worse)
Severity of dry nose | in the first 24 hours
  Patient reported outcome criteria (PRO); min=0;max=100(worse)
Severity of feeling of gastric distension | in the first 24 hours
  Patient reported outcome criteria (PRO); min=0;max=100(worse)
Constipation | in the first 48 hours
  Constipation (PRO); min=0;max=100(worse)
Nausea | in the first 48 hours
  Patient reported outcome criteria (PRO) ;min=0;max=100(worse)
Nurses' adherence to the protocol | in the first 24 hours
  Nurses' adherence to the protocol (questionnaire)
Nurses' satisfaction with the protocol | in the first 24 hours
  Nurses' satisfaction with the protocol (questionnaire)
Number of non invasive ventilation sessions | in the first 24 hours
  Number of non invasive ventilation sessions
Total duration of non invasive ventilation | in the first 24 hours
  Total duration of non invasive ventilation (number of hours)
Tolerance of non invasive ventilation | in the first 24 hours
  Tolerance of non invasive ventilation (PRO) ;min=0;max=100(worse)
Duration of HFNCO (high-flow nasal canula oxygenation) | in the first 24 hours
  Duration of HFNCO (number of hours)
Tolerance of HFNCO(high-flow nasal canula oxygenation) | in the first 24 hours
  Tolerance of HFNCO : number of adverses events
Duration of standard oxygen | in the first 24 hours
  Duration of standard oxygen (number of hours)
Tolerance of standard oxygen | in the first 24 hours
  Tolerance of standard oxygen : number of adverses events
Any adverse or serious event occurring | within the first 48 hours
  Any adverse or serious event occurring

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DEMOULE, PH, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Deleris R, Bureau C, Lebbah S, Decavele M, Dres M, Mayaux J, Similowski T, Dechartres A, Demoule A. Low dose of morphine to relieve dyspnea in acute respiratory failure: the OpiDys double-blind randomized controlled trial. Respir Res. 2024 Jul 16;25(1):280. doi: 10.1186/s12931-024-02867-2. PMID 39014448
- [Derived] Demoule A, Deleris R, Bureau C, Lebbah S, Decavele M, Dres M, Similowski T, Dechartres A. Low dose of morphine to relieve dyspnea in acute respiratory failure (OpiDys): protocol for a double-blind randomized controlled study. Trials. 2022 Sep 30;23(1):828. doi: 10.1186/s13063-022-06754-3. PMID 36175968